CLINICAL TRIAL: NCT04520412
Title: A Phase 3, Multi-center, Randomized, Double-blind, Parallel-group, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Sodium Oligomannate (GV-971) in Treatment of Mild to Moderate Alzheimer's Disease (GREEN MEMORY: GREen Valley 971 EvaluatioN Memory)
Brief Title: A Study of Sodium Oligomannate (GV-971) in Participants With Mild to Moderate Alzheimer's Disease
Acronym: GREEN MEMORY
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The quality of study was seriously affected by the COVID-19, so it was decided to suspend the trial and restart it at the right time.
Sponsor: Green Valley (Shanghai) Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GV971-007
Record Dates: First submitted 2020-08-11; First posted 2020-08-20 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — GV-971

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GV-971 (Experimental)
  Interventions: Drug: GV-971
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GV-971 — Administered PO
  Arms: GV-971
Drug: Placebo — Administered PO
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of GV-971 in mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate AD per NIA-AA.
* History of cognitive and functional decline over at least 1 year.
* MMSE scores between 11 and 24 (inclusive) at baseline.
* Brain MRI scan show the highest possibility of AD.
* Have a study partner/caregiver.

Exclusion Criteria:

* Diagnosis of a dementia-related central nervous system disease other than AD.
* Major structural brain disease as judged by MRI.
* A resting heart rate of < 50 beats per minute (bpm) after 5 minutes of rest in sitting or supine position.
* Major medical illness or unstable medical condition within 6 months of screening.
* Concomitant use of AChEIs and/or memantine within 30 days before first MMSE score, and during the study.
* Inadequate hepatic function.
* Inadequate organ and marrow function.
* ECG clinically significant abnormalities.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2046 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the ADAS-cog/11 score | Baseline, 48 weeks and 52 weeks
  Change from baseline in Alzheimer's Disease Assessments Scale - cognitive (ADAS-cog/11) scale total score. The total score of ADAS-cog/11 is 0-70, with higher scores mean a worse outcome.
Change from baseline in the ADCS-CGIC score | Baseline, 48 weeks and 52 weeks
  Change from baseline on Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) scale total score. The total score of ADCS-CGIC is 1-7, with higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from baseline in NPI score | Baseline, 36 Weeks, 52 Weeks
  Change from baseline in Neuropsychiatric Inventory (NPI) score. The total score of NPI is 0-144, with higher scores mean a worse outcome.
Change from baseline in MMSE score | Baseline, 52 Weeks
  Change from baseline in Mini Mental State Examination (MMSE) score. The total score of MMSE is 0-30, with higher scores mean a better outcome.
Change from baseline in ADCS-ADL23 score | Baseline, 36 Weeks, 52 Weeks
  Change from baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living; 23-item Scale (ADCS-ADL23) score. The total score of ADCS-ADL23 is 0-78, with higher scores mean a better outcome.
Change from baseline in NPI caregiver items | Baseline, 52 Weeks
  Change from baseline in Neuropsychiatric Inventory (NPI) caregiver items . The total score of NPI caregiver items is 0-60, with higher scores mean a worse outcome.
Change from baseline in ZBI score | Baseline, 52 Weeks
  Change from baseline in Zarit Burden Interview (ZBI) score. The total score of ZBI is 0-88, with higher scores mean a worse outcome.
Assess the efficacy of GV-971 throughout the OLE period | Baseline, 52 Weeks, 78 Weeks
  Change from baseline in Alzheimer's Disease Assessments Scale - cognitive (ADAS-cog/11) scale total score. The total score of ADAS-cog/11 is 0-70, with higher scores mean a worse outcome.
Assess the efficacy of GV-971 throughout the OLE period | Baseline, 52 Weeks, 78 Weeks
  Change from baseline on Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) scale total score. The total score of ADCS-CGIC is 1-7, with higher scores mean a worse outcome.

OTHER OUTCOMES:
Evaluate the population PK | Baseline, 12 Weeks, 24 Weeks, 52 Weeks
  Determine serum levels of GV-971 in population PK
Evaluate the effect of GV-971 on brain structure neurodegeneration | Baseline, 52 Weeks
  Changes from baseline in volumetric magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Ph D, Study Director — Green Valley (Shanghai) Pharmaceuticals Co., Ltd.
Locations (171):
- United States (67):
  - Cognitive Clinical Trials, LLC, Gilbert, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Banner Alzheimer's Institute, Tucson, Arizona
  - Irvine Clinical Research, Irvine, California
  - Sunwise Clinical Research, Lafayette, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Research Network, Inc, San Diego, California
  - Pacific Research Network, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Schuster Med Research Institute, Sherman Oaks, California
  - JEM Research LLC, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Finlay Medical Research Corp, Greenacres City, Florida
  - Velocity Clinical Research, Hallandale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Charter Research, LLC, Lady Lake, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - ClinCloud, LLC, Maitland, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Suncoast Clinical Research Inc., New Port Richey, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Synexus Clinical Research, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Quantum Lab CNS Clinical Research, Pompano Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Synexus The Villages, The Villages, Florida
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Alliance Multispecialty Research, Wichita, Kansas
  - Activmed Practices&Research, Lawrence, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Barnes-Jewish Hospital IDS, St Louis, Missouri
  - University of Nebraska Medical Center-Hematology/Oncology Section, Omaha, Nebraska
  - Cognitive Clinical Trials, LLC, Omaha, Nebraska
  - Altea Research Institute, Las Vegas, Las Vegas, Nevada
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - The Cognitive Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ, PC, Toms River, New Jersey
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - UBMD Neurology, Buffalo, New York
  - Clarity Clinical Research, East Syracuse, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Behavioral Health Research Center, Charlotte, North Carolina
  - AMC Research, LLC, Charlotte, North Carolina
  - Guilford Neurologic Associate, Greensboro, North Carolina
  - Insight Clinical Trials LLC, Beachwood, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Neuroscience, LLC, Westerville, Ohio
  - Summit Research Network(Oregon)Inc., Portland, Oregon
  - Oregon Health&Science Universty, Portland, Oregon
  - Oregon Neurology Associates, Springfield, Oregon
  - Abington Neurological Associates, LTD, Abington, Pennsylvania
  - SCarolina Institute Brain Health, Charleston, South Carolina
  - Kerwin Research Center, Dallas, Texas
  - Huston Methodist Hospital, Houston, Texas
  - Clinical Trials of Texas; Inc, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Cognition Health, Fairfax, Virginia
  - University Washington MedCentre, Seattle, Washington
- Australia (4):
  - Hornsby Ku-ring-gai Hospital, Hornsby, New South Wales
  - KaRa MINDS, Macquarie Park, New South Wales
  - Austin Health - Heidelberg Repatriation Hospital, Melbourne, Victoria
  - Alzheimer's Research Foundation, Nedlands, Western Australia
- Canada (17):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - The Medical Arts Health Research Group, Kamloops, British Columbia
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - MedicalArtsHealth Research Grp, Kelowna, British Columbia
  - MedicalArtsHealth Research Grp, Penticton, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Medical Arts Health Research Grp, West Vancouver, British Columbia
  - True North Clinical Research Inc, Halifax, Nova Scotia
  - True North Clinical Research, New Minas, Nova Scotia
  - Recherches Neuro-Hippocampe Inc., d/b/a Ottawa Memory Clinic, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Clinique Memoire Outaouais, Gatineau, Quebec
  - Q & T Research Sherbrooke Inc, Sherbrooke, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
  - Douglas Hospital Research Centre, Verdun, Quebec
  - ALPHA Recherche Clinique, Québec
- China (44):
  - 1st Hospital of Anhui MU, Hefei, Anhui
  - Peking Union Hospital, Beijing, Beijing Municipality
  - Peking University 1st Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tong Ren Hospital, Beijing, Beijing Municipality
  - 1st Hospital of Chongqing MU, Chongqing, Chongqing Municipality
  - Fujian Union Hospital, Fuzhou, Fujian
  - 1st Hospital of Fujian MU, Fuzhou, Fujian
  - Zhongshan Hospital Xiamen U, Xiamen, Fujian
  - 1st Hospital of Guangzhou MU, Guangzhou, Guangdong
  - Guangzhou 1st People's Hospital, Guangzhou, Guangdong
  - 2nd Hospital of Guangzhou MU, Guangzhou, Guangdong
  - 2nd Hospital Zhongshan University, Guangzhou, Guangdong
  - Kangning Hospital of Shenzhen, Shenzhen, Guangdong
  - 1st Hospital of Hebei MU, Shijiazhuang, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - Xiangya Hospital, Changsha, Hunan
  - Yueyang 1st People's Hospital, Yueyang, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhong Da Hospital, Nanjing, Jiangsu
  - 2nd Hospital Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Hospital, Nanchang, Jiangxi
  - 1st Hospital Jilin University, Changchun, Jilin
  - General Hospital of Ningxia MU, Yinchuan, Ningxia
  - Tang Du Hospital, Xi'an, Shaanxi
  - Xi'an Mental Health Cente, Xi'an, Shaanxi
  - Qilu Hospital, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Huashan Hospital; Fudan U, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - 1st Hospital of Shanxi MU, Taiyuan, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - Tianjin MU General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - 1st Hospital of Kunming MU, Kunming, Yunnan
  - Zhejiang Provincial Hospital, Hangzhou, Zhejiang
  - 1st Hospital Zhejiang University, Hangzhou, Zhejiang
  - 1st Hospital of Wenzhou MU, Wenzhou, Zhejiang
- Czechia (6):
  - NeuropsychiatrieHK s.r.o., Hradec Králové
  - BRAIN-SOULTHERAPY s.r.o., Kladno
  - Neuroterapie KH s.r.o., Kutná Hora
  - Clintrial s.r.o., Prague
  - FORBELI s.r.o., Prague
  - Neuropsychiatrie s.r.o., Prague
- France (14):
  - Centred Investigation Clinique, Strasbourg, Bas Rhin
  - CHUTimone Adultes Service, Marseille, Bouches-du-Rhône
  - HOPITAL Gui de CHAULIAC, Montpellier, Cedex 5
  - Centre Memoire Ressources, Dijon, De Lattre de Tassigny
  - Groupe Hospitalier Pellegrin, Bordeaux, Gironde
  - Hopitaux Civils de Colmar, Colmar, Grand Est
  - Recherche Clinique Gerontopole, Toulouse, Haute Garonne
  - Pharmacie CHU de Rennes, Rennes, Ille Et Vilaine
  - CHU Tours-Hopital Bretonneau, Tonnerre, Indre Et Loire
  - CHU Nantes-Hopital Nord Laennec, Nantes, Loire Atlantique
  - CHU Reims-Hopital Maison Blanche, Reims, Marne
  - Neurologique Pierre Wertheimer, Bron, Rhone
  - Hopital des Charpennes, Villeurbanne, Rhone
  - CMRR Paris Nord, Paris
- Prince of Wales Hospital, Shatin, Hong Kong
- Netherlands (4):
  - VUmc Goederenontvangst, Amsterdam, Van Der Boechorststraat 6
  - Pharmacy Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Amphia Hospital Breda, Breda
  - Klinische Farmacie, Zwolle
- Poland (11):
  - Podlaskie Centrum Psychogeriatri, Bialystok
  - NZOZ Vitamed, Bydgoszcz
  - Wielospec. Poradnia Lekarska, Katowice
  - Nzoz Novo Med, Katowice
  - Specjalistyczne Gabinety Sp.zo.o, Krakow
  - NZOZ Neuromed MiMNastajSpp, Lublin
  - Medicome Sp z o o, Oświęcim
  - Solumed Centrum Medyczne, Poznan
  - Neuro Protect, Warsaw
  - Wrclawskie Cntrm Alzheimerowskie, Wroclaw
  - Wielospecjalistyczne Centrm Med, Zabrze
- Taiwan (3):
  - National Taiwan UniversityHosp, Taipei
  - Tri Service General Hospital, Taipei
  - Chang GungMemorial Hosp Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided